CLINICAL TRIAL: NCT04093739
Title: Post-market Clinical Follow-up Study of the G7 Freedom Constrained Neutral Liner and G7 Neutral +5mm Liner in Primary and Revision Total Hip Arthroplasty (Implants and Instrumentation)
Brief Title: MDR - G7 Neutral and G7 Freedom Constrained Neutral Acetabular Liners
Status: Withdrawn | Type: Observational
Why Stopped: Manufacturer decided not to proceed with study.
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: MDRG2017-89MS-53H
Record Dates: First submitted 2019-07-18; First posted 2019-09-18 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Hip Osteoarthritis; Hip Disease; Hip Fractures; Hip Injuries
MeSH Terms: conditions — Osteoarthritis, Hip; Hip Fractures; Hip Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- G7 Freedom Constrained Liners: Patients that have been implanted with a G7 Freedom Constrained liner to repair hip malfunction or disease.
  Interventions: Device: G7 Freedom Constrained Liners

INTERVENTIONS:
Device: G7 Freedom Constrained Liners — Patients that have been implanted with the G7 Freedom Constrained Liners to repair hip malfunction and/or disease.

SUMMARY:
The objective of this consecutive series PMCF study is to collect data confirming safety, performance and clinical benefits of the G7 Freedom Constrained Liners when used for primary and revision total hip arthroplasty (implants and instrumentation) at 5 years follow-up. Since G7 Acetabular Cup System has only been on the market since 2015, a prospective follow-up will be necessary to obtain data for the 5 year post-surgery time-point for each patient.

DETAILED DESCRIPTION:
The objective of this consecutive series PMCF study is to collect data confirming safety, performance and clinical benefits of the G7 Freedom Constrained Liners when used for primary and revision total hip arthroplasty (implants and instrumentation) at 5 years follow-up. Since G7 Acetabular Cup System has only been on the market since 2015, a prospective follow-up will be necessary to obtain data for the 5 year post-surgery time-point for each patient.

The primary objective is to confirm safety of the study products. This will be assessed by recording the incidence and frequency of revisions, complications, and adverse events. Relationship of the events to either implant or instrumentation should be specified.

The secondary objective is the assessment of performance and clinical benefits by analyzing recorded patient-reported clinical outcomes measures (PROMs).

ELIGIBILITY:
Inclusion Criteria:

* Patient must be 18 years of age or older and skeletally mature
* Patient must be willing and able to sign Institution Review Board (IRB) approved informed consent
* Noninflammatory degenerative joint disease including:
* Osteoarthritis
* Avascular necrosis
* Rheumatoid arthritis
* Correction of functional deformity
* Treatment of non-union, femoral neck fracture, and trochanteric fractures of the proximal femur with head involvement, unmanageable by other -techniques
* High risk of dislocation due to:
* History of prior dislocation
* Bone loss
* Joint or soft tissue laxity
* Neuromuscular disease
* Intraoperative instability
* Revision procedures where other treatment or devices have failed

Exclusion Criteria:

* Off-label use
* Infection and/or distant foci of infections which may spread to the implant site
* Sepsis
* Osteomyelitis
* Uncooperative patient or patient with neurologic disorders who are incapable of following directions
* Osteoporosis
* Metabolic disorders which may impair bone formation
* Osteomalacia
* Rapid joint destruction, marked bone loss or bone resorption apparent on roentgenogram
* Vascular insufficiency, muscular atrophy or neuromuscular disease
* Patient is known to be pregnant or nursing
* Patient is a prisoner
* Patient is a known alcohol or drug abuser
* Patient has a psychiatric illness or cognitive deficit that will not allow for proper informed consent
* Patient is unwilling to sign an informed consent

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This will include a consecutive series of subjects implanted with the G7 Freedom Constrained Liners in primary and revision total hip arthroplasty according to the approved
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-04 (Estimated); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Device Safety assessed through the frequency and incidence of revisions, complications and adverse events | Out to five years
  The primary objective is to confirm safety of the study products. This will be assessed by recording the incidence and frequency of revisions, complications, and adverse events. Relationship of the events to either implant or instrumentation should be specified.

SECONDARY OUTCOMES:
Device Performance and Benefits evaluated through the Oxford Hip Score | Out to five years
  The OHS is a patient completed 12 question evaluation. Each item is scored from 1 to 5, with 1 representing best outcome/least symptoms and 5 representing worst outcome/most symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Erin Osborn, Study Director — Zimmer Biomet

IPD SHARING:
Plan to Share IPD: No